CLINICAL TRIAL: NCT02080312
Title: Magnetic Resonance Imaging Evaluation of Inner Ear Pathology Using Intra-Tympanic Contrast Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Society of Head and Neck Radiology (Unknown)
Responsible Party: Principal Investigator, Julie Bykowski, MD, Assistant Professor, Radiology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 120004; 115,342 (Other: FDA)
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Meniere's Disease
Keywords: Meniere's disease; endolymphatic hydrops
MeSH Terms: conditions — Meniere Disease; Endolymphatic Hydrops | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intratympanic injection (Experimental): Magnevist (gadopentetate dimeglumine, Bayer Health Care) will be diluted eightfold with sterile saline (1:7 v/v) in a 1 ml syringe and injected intra-tympanically with a 23-25g needle up to 0.4 ml or less if contrast reflux is noted under direct visualization. Anesthesia with topical phenol is available for this procedure.
  Interventions: Drug: Magnevist (gadopentetate dimeglumine)

INTERVENTIONS:
Drug: Magnevist (gadopentetate dimeglumine)

SUMMARY:
This is a pilot study of patients with clinical symptoms of Ménière's disease using injection of diluted magnetic resonance imaging (MRI) contrast agent into the ear to evaluate inner ear structures.

The goal is to reproduce imaging findings described by non-United States (US) institutions, improve on image quality with decreased scan time and evaluate the dynamics of the contrast movement into the inner ear structures.

DETAILED DESCRIPTION:
Participants will be scheduled for study sessions on 2 consecutive days to include consent, baseline audiometric evaluation, intra-tympanic contrast administration, serial MR imaging, and follow-up audiometry evaluation in the injected ear.

Participants over 59 years old or who have medical conditions will have a blood test to check kidney function to ensure they can safely receive the contrast.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and clinical exam consistent with Ménière's disease
* Ability to undergo MR exam
* Interest in participating in this study
* Ability to provide informed consent

Exclusion Criteria:

* Children (under age 18),
* Contraindication to MR imaging (see attached UCSD MR Screening Form)
* Claustrophobia precluding MR exam without sedation
* Contraindication to receiving intravenous gadolinium-based contrast agent (see attached UCSD Contrast Policy)
* Patients who are pregnant or breast feeding (intravenous contrast agents are Category C)
* Contraindication to osmotic challenge (congestive heart failure, renal failure, hepatic failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Health System, San Diego, California, United States

REFERENCES:
- [Result] Bykowski J, Harris JP, Miller M, Du J, Mafee MF. Intratympanic Contrast in the Evaluation of Meniere Disease: Understanding the Limits. AJNR Am J Neuroradiol. 2015 Jul;36(7):1326-32. doi: 10.3174/ajnr.A4277. Epub 2015 Mar 26. PMID 25814661

RESULTS

PARTICIPANT FLOW:
Groups:
- Intratympanic Injection: Magnevist (gadopentetate dimeglumine, Bayer Health Care) will be diluted eightfold with sterile saline (1:7 v/v) in a 1 ml syringe and injected intra-tympanically with a 23-25g needle up to 0.4 ml or less if contrast reflux is noted under direct visualization. Anesthesia with topical phenol is available for this procedure.
  Magnevist (gadopentetate dimeglumine)
Period: Overall Study
Arm/Group | Intratympanic Injection
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intratympanic Injection
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Vestibular "Endolymphatic Hydrops (EH)"
Description: The relative volume of the non-enhancing endolymphatic space was visually assessed relative to the enhancing perilymphatic space on delayed post-IT contrast FLAIR MRI sequences and characterized as <34%, 34-50% or >50% of endolymphatic/perilymphatic volume.
Time Frame: 24 hours post injection
Measure: Number; unit: participants
Arm/Group | Intratympanic Injection
Number analyzed (Participants) | 6
participants
  Vestibular EH < 34% | 0
  Vestibular EH 34-50% | 4
  Vestibular EH >50% | 2

2. Primary Outcome: Cochlear "Endolymphatic Hydrops (EH)"
Description: The relative volume of the scala media of the basal turn of the cochlea (non-enhancing endolymph) was visually assessed relative to the scala tympani and scala vestibuli (enhancing perilymph) on delayed post-IT contrast FLAIR MRI sequences. Cases were characterized as: No Cochlear EH (no perceptible distention of the scala media), Cochlear EH (perceptible distention of the scala media), or Absent enhancement (no contrast in the cochlear perilymph)
Time Frame: 24 hours post injection
Measure: Number; unit: participants
Arm/Group | Intratympanic Injection
Number analyzed (Participants) | 6
participants
  No Cochlear EH | 0
  Cochlear EH | 6
  Absent enhancement | 0

3. Secondary Outcome: Extension of Contrast From Perilymph to CSF
Description: The fundus of the internal auditory canal (IAC) was visually inspected to determine if there was conspicuous, subtle, or no enhancement extending in the setting of prior IT contrast injection, indicating permeability of the cochlear modiolus.
Time Frame: 24 hours post injection
Measure: Number; unit: participants
Arm/Group | Intratympanic Injection
Number analyzed (Participants) | 6
participants
  Conspicuous enhancement in IAC | 1
  Subtle enhancement in IAC | 2
  No enhancement in IAC | 3

ADVERSE EVENTS:
Arm/Group | Intratympanic Injection
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No